CLINICAL TRIAL: NCT03860636
Title: The Prognostic Accuracy of Within Cycle, Pre-embryo Transfer, Ultrasound Endometrial Patterns, to Predict Implantation During Assisted Reproduction
Brief Title: The Accuracy of Endometrial Ultrasound to Predict Implantation
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Nick Raine Fenning, Chief Investigator, University of Nottingham
Other Study IDs: REC 87-1808
Record Dates: First submitted 2018-11-02; First posted 2019-03-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Infertility, Subfertility
Keywords: In Vitro Fertilisation (IVF); Intra Cytoplasmic Injection (ICSI); Endometrial Pattern; Ultrasound
MeSH Terms: conditions — Infertility | interventions — Hematologic Tests; Echocardiography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for progesterone and estradiol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fresh Embryo Transfer: Women will be invited to attend and have transvaginal ultrasound scans (TVUS) and blood tests at three different points during their treatments.
  * The day they receive their HCG trigger,
  * The day of transvaginal oocyte retrieval (TVOR) and
  * The day of embryo transfer (ET).
  Interventions: Diagnostic Test: Endometrial Pattern on Ultrasound at ET; Diagnostic Test: Endometrial Pattern on Ultrasound at HCG; Diagnostic Test: Endometrial Pattern on Ultrasound at TVOR; Diagnostic Test: Endometrial thickness at HCG; Diagnostic Test: Endometrial thickness at TVOR; Diagnostic Test: Endometrial thickness at ET; Diagnostic Test: Endometrial volume at HCG; Diagnostic Test: Endometrial volume at TVOR; Diagnostic Test: Endometrial volume at ET; Diagnostic Test: Blood test for progesterone at HCG; Diagnostic Test: Blood test for progesterone at TVOR; Diagnostic Test: Blood test for progesterone at ET; Diagnostic Test: Blood test for estradiol at HCG; Diagnostic Test: Blood test for estradiol at TVOR; Diagnostic Test: Blood test for estradiol at ET; Diagnostic Test: Endometrial blood flow (doppler) at HCG; Diagnostic Test: Endometrial blood flow (doppler) at TVOR; Diagnostic Test: Endometrial blood flow (doppler) at ET; Diagnostic Test: Contractility at embryo transfer on a subgroup of participants; Diagnostic Test: Change in endometrial pattern between HCG and ET
- Frozen Embryo Transfer: Women will be invited to attend and have transvaginal ultrasound scans (TVUS) and blood tests at two different points during their treatments.
  * The day we coordinate with embryologist (day of progesterone +/-1)
  * The day of embryo transfer (ET).
  Interventions: Diagnostic Test: Endometrial Pattern on Ultrasound at ET; Diagnostic Test: Endometrial Pattern on Ultrasound at co-ordination scan; Diagnostic Test: Endometrial thickness at ET; Diagnostic Test: Endometrial thickness at coordination scan; Diagnostic Test: Endometrial volume at ET; Diagnostic Test: Endometrial volume at coordination scan; Diagnostic Test: Blood test for progesterone at ET; Diagnostic Test: Blood test for progesterone at coordination scan; Diagnostic Test: Change in endometrial pattern between TVOR and ET; Diagnostic Test: Blood test for estradiol at ET; Diagnostic Test: Blood test for estradiol at coordination scan; Diagnostic Test: Endometrial blood flow (doppler) at ET; Diagnostic Test: Endometrial blood flow (doppler) at coordination scan; Diagnostic Test: Contractility at embryo transfer on a subgroup of participants; Diagnostic Test: Change in endometrial pattern between coordination scan and ET

INTERVENTIONS:
Diagnostic Test: Endometrial Pattern on Ultrasound at ET — Ultrasound scan
Diagnostic Test: Endometrial Pattern on Ultrasound at HCG — Ultrasound
  Groups: Fresh Embryo Transfer
Diagnostic Test: Endometrial Pattern on Ultrasound at TVOR — Ultrasound
  Groups: Fresh Embryo Transfer
Diagnostic Test: Endometrial Pattern on Ultrasound at co-ordination scan — Ultrasound
  Groups: Frozen Embryo Transfer
Diagnostic Test: Endometrial thickness at HCG — Ultrasound
  Groups: Fresh Embryo Transfer
Diagnostic Test: Endometrial thickness at TVOR — Ultrasound
  Groups: Fresh Embryo Transfer
Diagnostic Test: Endometrial thickness at ET — Ultrasound scan
Diagnostic Test: Endometrial thickness at coordination scan — Ultrasound scan
  Groups: Frozen Embryo Transfer
Diagnostic Test: Endometrial volume at HCG — Ultrasound scan
  Groups: Fresh Embryo Transfer
Diagnostic Test: Endometrial volume at TVOR — Ultrasound scan
  Groups: Fresh Embryo Transfer
Diagnostic Test: Endometrial volume at ET — Ultrasound scan
Diagnostic Test: Endometrial volume at coordination scan — Ultrasound scan
  Groups: Frozen Embryo Transfer
Diagnostic Test: Blood test for progesterone at HCG — Blood test
  Groups: Fresh Embryo Transfer
Diagnostic Test: Blood test for progesterone at TVOR — Blood test
  Groups: Fresh Embryo Transfer
Diagnostic Test: Blood test for progesterone at ET — Blood test
Diagnostic Test: Blood test for progesterone at coordination scan — Blood test
  Groups: Frozen Embryo Transfer
Diagnostic Test: Change in endometrial pattern between TVOR and ET — Ultrasound scan
  Groups: Frozen Embryo Transfer
Diagnostic Test: Blood test for estradiol at HCG — Blood test
  Groups: Fresh Embryo Transfer
Diagnostic Test: Blood test for estradiol at TVOR — Blood test
  Groups: Fresh Embryo Transfer
Diagnostic Test: Blood test for estradiol at ET — Blood test
Diagnostic Test: Blood test for estradiol at coordination scan — Blood test
  Groups: Frozen Embryo Transfer
Diagnostic Test: Endometrial blood flow (doppler) at HCG — Ultrasound scan
  Groups: Fresh Embryo Transfer
Diagnostic Test: Endometrial blood flow (doppler) at TVOR — Ultrasound scan
  Groups: Fresh Embryo Transfer
Diagnostic Test: Endometrial blood flow (doppler) at ET — Ultrasound scan
Diagnostic Test: Endometrial blood flow (doppler) at coordination scan — Ultrasound scan
  Groups: Frozen Embryo Transfer
Diagnostic Test: Contractility at embryo transfer on a subgroup of participants — Ultrasound scan
Diagnostic Test: Change in endometrial pattern between coordination scan and ET — Ultrasound scan
  Groups: Frozen Embryo Transfer
Diagnostic Test: Change in endometrial pattern between HCG and ET — Ultrasound scan
  Groups: Fresh Embryo Transfer

SUMMARY:
To measure the accuracy of different ultrasound endometrial patterns to predict successful embryo implantation during assisted conception; in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI).

DETAILED DESCRIPTION:
Ultrasound appearance of the endometrium may predict successful implantation in assisted conception, but studies have yielded conflicting results.

The explanation may be different timing of, and classification systems for, the scan, different treatment protocols, and different definitions of success. Also scan quality has improved over time.

This is a prospective study looking at the endometrial pattern as a predictor of IVF/ICSI outcome, adjusting for embryo quality, ease of transfer, and fresh or frozen cycles. The study will focus on good quality single embryo transfer at the blastocyst stage. Other endometrial ultrasound parameters such as thickness, volume and Doppler will also be measured. Reliability studies will also be conducted to assess and account for inter- and intra-observer variation.

200 women will be recruited. They will include approximately 100 undergoing fresh and 100 undergoing frozen embryo transfer. There will be no change to routine clinical care. A single operator will analyse all ultrasound images to reduce inter-observer variation. When there is uncertainty about the pattern the chief investigator will be consulted to reach an agreement.

ELIGIBILITY:
Inclusion Criteria:

* Female undergoing in vitro fertilisation or intracytoplasmic sperm injection (IVF/ICSI)
* Own or donated eggs
* Informed consent

Exclusion Criteria:

* Known pathology affecting the endometrial cavity (polyp, submucosal fibroid)
* Septate uterus or more complex uterine abnormality.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Women who are having in vitro fertilisation or intracytoplasmic sperm injection where a clear image of endometrial pattern can be obtained. In cases where we can't obtain a clear endometrial pattern due to pathology or uterine position, we will exclude these cases from analysis. In cases of failure of fertilisation where no embryo is available for transfer these cases will be excluded from analysis.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Number of clinical pregnancies | Within 12 weeks after embryo transfer (usually scan performed at 6-7 weeks gestation)
  Intrauterine pregnancy with fetal heart detected on ultrasound arising from the treatment cycle

SECONDARY OUTCOMES:
Number of ectopic pregnancies | Within 10 weeks after embryo transfer
  Ectopic pregnancy resulting from the treatment cycle
Number of biochemical pregnancies | Within 6 weeks after embryo tranfer
  Biochemical pregnancy resulting from the treatment cycle
Number of miscarriages | Within 12 weeks after embryo transfer
  Miscarriage resulting from the treatment cycle
Number of live birth | Within one year after embryo transfer
  Live birth resulting from the treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Raine-Fenning, MRCOG PhD, Principal Investigator — University of Nottingham, Nurture Fertility Director
Locations (1):
- Nurture Fertility, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided